CLINICAL TRIAL: NCT01464476
Title: Phase 3 Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Effects of Once Daily Oral Doses of 75 mg Azimilide Dihydrochloride on the Incidence of Cardiovascular Hospitalizations/Emergency Department Visits or Cardiovascular Death in Patients With an Implantable Cardioverter Defibrillator
Brief Title: Efficacy and Safety Study of Azimilide on the Incidence of Cardiovascular Hospitalizations/Emergency Department Visits or Cardiovascular Death in Patients With an Implantable Cardioverter Defibrillator (ICD) (SHIELD-2)
Acronym: SHIELD-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AZM-MD-302
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases | interventions — azimilide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azimilide (Experimental): Azimilide 75 mg film coated tablets
  Interventions: Drug: Azimilide Dihydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azimilide Dihydrochloride — Azimilide 75 mg. Once daily, oral administration
  Arms: Azimilide
Drug: Placebo — Dose-matched placebo. Once daily, oral administration
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of Azimilide on the incidence of cardiovascular hospitalizations, cardiovascular emergency department visits or cardiovascular death in patients with Implantable Cardioverter Defibrillators (ICDs)

ELIGIBILITY:
Inclusion Criteria:

* Have an ICD implanted and a history of ventricular tachycardia, ventricular fibrillation, or an appropriate ICD therapy.
* Have a left ventricular ejection fraction <= 0.40

Exclusion Criteria:

* Have New York Heart Association (NYHA) Class IV Congestive Heart Failure (CHF) or have decompensated CHF at the time of randomization;
* Have unstable angina pectoris or a myocardial infarction within 30 days of randomization;
* Have a history of Torsade de Pointes or heart transplantation
* Have chronic atrial fibrillation or atrial fibrillation/flutter, that is not adequately rate controlled in the judgment of the Investigator, at screening;
* Are currently taking systemic Class I or other Class III antiarrhythmic drugs
* Are currently taking systemic drugs that prolong the QT interval
* If female, are currently pregnant or breast feeding, or plan to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Time to first cardiovascular event | 365 days
  Time to first unplanned cardiovascular hospitalization, unplanned cardiovascular emergency department visit, or cardiovascular death in patients with an Implantable Cardioverter Defibrillator (ICD)

SECONDARY OUTCOMES:
Time to first all-cause shock by the ICD | 365 days
  Time to first all-cause shock initiated by the Implantable Cardioverter Defibrillator
Time to first unplanned physician-office visit. | 365 days
  Time to the first unplanned physician-office visit.

CONTACTS AND LOCATIONS:
Overall Officials: David B Bharucha, MD, PhD, Study Director — Forest Laboratories
Locations (138):
- United States (83):
  - Forest Investigative Site 053, Birmingham, Alabama
  - Forest Investigative Site 048, Huntsville, Alabama
  - Forest Investigative Site 013, Phoenix, Arizona
  - Forest Investigative Site 110, Los Angeles, California
  - Forest Investigative Site 022, Merced, California
  - Forest Investigative Site 060, Colorado Springs, Colorado
  - Forest Investigative Site 090, Littleton, Colorado
  - Forest Investigative Site 041, Newark, Delaware
  - Forest Investigative Site 113, Hollywood, Florida
  - Forest Investigative Site 010, Jacksonville, Florida
  - Forest Investigative Site 035, Lakeland, Florida
  - Forest Investigative Site 044, Port Charlotte, Florida
  - Forest Investigative Site 062, Rockledge, Florida
  - Forest Investigative Site 082, Safety Harbor, Florida
  - Forest Investigative Site 006, Zephyrhills, Florida
  - Forest Investigative Site 123, Augusta, Georgia
  - Forest Investigative Site 092, Boise, Idaho
  - Forest Investigative Site 012, Bloomington, Indiana
  - Forest Investigative Site 068, Indianapolis, Indiana
  - Forest Investigative Site 087, South Bend, Indiana
  - Forest Investigative Site 063, Houma, Louisiana
  - Forest Investigative Site 050, Auburn, Maine
  - Forest Investigative Site 030, Baltimore, Maryland
  - Forest Investigative Site 058, Baltimore, Maryland
  - Forest Investigative Site 052, Lanham, Maryland
  - Forest Investigative Site 118, Silver Spring, Maryland
  - Forest Investigative Site 015, Boston, Massachusetts
  - Forest Investigative Site 091, Brighton, Massachusetts
  - Forest Investigative Site 020, Saginaw, Michigan
  - Forest Investigative Site 085, Southfield, Michigan
  - Forest Investigative Site 079, Troy, Michigan
  - Forest Investigative Site 034, Ypsilanti, Michigan
  - Forest Investigative Site 121, Tupelo, Mississippi
  - Forest Investigative Site 088, St Louis, Missouri
  - Forest Investigative Site 100, St Louis, Missouri
  - Forest Investigative Site 055, Englewood, New Jersey
  - Forest Investigative Site 059, Ridgewood, New Jersey
  - Forest Investigative Site 106, Warren Township, New Jersey
  - Forest Investigative Site 112, Albuquerque, New Mexico
  - Forest Investigative Site 018, Albany, New York
  - Forest Investigative Site 069, Albany, New York
  - Forest Investigative Site 045, New York, New York
  - Forest Investigative Site 122, New York, New York
  - Forest Investigative Site 075, Williamsville, New York
  - Forest Investigative Site 089, Chapel Hill, North Carolina
  - Forest Investigative Site 116, Greensboro, North Carolina
  - Forest Investigative Site 070, Canton, Ohio
  - Forest Investigative Site 064, Cincinnati, Ohio
  - Forest Investigative Site 124, Cincinnati, Ohio
  - Forest Investigative Site 043, Columbus, Ohio
  - Forest Investigative Site 083, Kettering, Ohio
  - Forest Investigative Site 109, Toledo, Ohio
  - Forest Investigative Site 119, Oklahoma City, Oklahoma
  - Forest Investigative Site 003, Tulsa, Oklahoma
  - Forest Investigative Site 056, Camp Hill, Pennsylvania
  - Forest Investigative Site 081, Erie, Pennsylvania
  - Forest Investigative Site 008, Erie, Pennsylvania
  - Forest Investigative Site 024, Hershey, Pennsylvania
  - Forest Investigative Site 095, Philadelphia, Pennsylvania
  - Forest Investigative Site 005, Wilkes-Barre, Pennsylvania
  - Forest Investigative Site 107, Yardley, Pennsylvania
  - Forest Investigative Site 046, York, Pennsylvania
  - Forest Investigative Site 084, Providence, Rhode Island
  - Forest Investigative Site 066, Florence, South Carolina
  - Forest Investigative Site 073, Greenville, South Carolina
  - Forest Investigative Site 014, Rapid City, South Dakota
  - Forest Investigative Site 094, Sioux Falls, South Dakota
  - Forest Investigative Site 029, Corpus Christi, Texas
  - Forest Investigative Site 028, Dallas, Texas
  - Forest Investigative Site 007, Fort Worth, Texas
  - Forest Investigative Site 111, Fort Worth, Texas
  - Forest Investigative Site 125, Houston, Texas
  - Forest Investigative Site 076, Houston, Texas
  - Forest Investigative Site 074, San Antonio, Texas
  - Forest Investigative Site 016, Chesapeake, Virginia
  - Forest Investigative Site 004, Falls Church, Virginia
  - Forest Investigative Site 117, Lynchburg, Virginia
  - Forest Investigative Site 065, Newport News, Virginia
  - Forest Investigative Site 072, Richmond, Virginia
  - Forest Investigative Site 023, Roanoke, Virginia
  - Forest Investigative Site 071, Green Bay, Wisconsin
  - Forest Investigative Site 042, Madison, Wisconsin
  - Forest Investigative Site 049, Milwaukee, Wisconsin
- Belgium (5):
  - Forest Investigative Site 302, Bruges
  - Forest Investigative Site 303, Charleroi
  - Forest Investigative Site 300, Leuven
  - Forest Investigative Site 304, Liège
  - Forest Investigative Site 301, Yvoir
- Canada (11):
  - Forest Investigative Site 264, Edmonton, Alberta
  - Forest Investigative Site 269, Vancouver, British Columbia
  - Forest Investigative Site 252, Victoria, British Columbia
  - Forest Investigative Site 267, Hamilton, Ontario
  - Forest Investigative Site 253, Kingston, Ontario
  - Forest Investigative Site 259, Toronto, Ontario
  - Forest Investigative Site 263, Toronto, Ontario
  - Forest Investigative Site 254, Montreal, Quebec
  - Forest Investigative Site 250, Montreal, Quebec
  - Forest Investigative Site 270, Sherbrooke, Quebec
  - Forest Investigative Site 262, Saskatoon, Saskatchewan
- Czechia (5):
  - Forest Investigative Site 750, Brno
  - Forest Investigative Site 753, České Budějovice
  - Forest Investigative Site 751, Olomouc
  - Forest Investigative Site 754, Prague
  - Forest Investigative Site 752, Sokolska
- Denmark (5):
  - Forest Investigative Site 852, Aalborg
  - Forest Investigative Site 850, Copenhagen
  - Forest Investigative Site 854, Esbjerg
  - Forest Investigative Site 853, Hellerup
  - Forest Investigative Site 851, Odense
- France (5):
  - Forest Investigative Site 353, Grenoble
  - Forest Investigative Site 354, Lille
  - Forest Investigative Site 350, Montpellier
  - Forest Investigative Site 358, Nantes
  - Forest Investigative Site 357, Pessac
- Germany (5):
  - Forest Investigative Site 405, Berlin
  - Forest Investigative Site 402, Göttingen
  - Forest Investigative Site 410, Heidelberg
  - Forest Investigative Site 406, Ludwigshafen
  - Forest Investigative Site 401, Mannheim
- Israel (4):
  - Forest Investigative Site 450, Ashkelon
  - Forest Investigative Site 453, Jerusalem
  - Forest Investigative Site 452, Tel Aviv
  - Forest Investigative Site 451, Tel Litwinsky
- Italy (2):
  - Forest Investigative Site 504, Ancona
  - Forest Investigative Site 502, Catania
- Netherlands (3):
  - Forest Investigative Site 552, Breda
  - Forest Investigative Site 550, Eindhoven
  - Forest Investigative Site 555, Zwolle
- Poland (2):
  - Forest Investigative Site 706, Gdansk
  - Forest Investigative Site 705, Gdynia
- Spain (2):
  - Forest Investigative Site 604, Barcelona
  - Forest Investigative Site 601, Málaga
- Sweden (6):
  - Forest Investigative Site 800, Lund
  - Forest Investigative Site 805, Örebro
  - Forest Investigative Site 804, Stockholm
  - Forest Investigative Site 802, Stockholm
  - Forest Investigative Site 801, Uppsala
  - Forest Investigative Site 803, Västerås